CLINICAL TRIAL: NCT07076069
Title: The Effect of Multimodal Pain Regimen on Use of Narcotics After Rotator Cuff Tear Repair
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-14249
Record Dates: First submitted 2025-07-13; First posted 2025-07-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Repairs; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Before surgeries, patients will be assigned to one of the two arms in a block randomization fashion in a 1:1 ratio. A block randomization scheme with a block size of 6 will be generated and maintained by the study statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Pain Regimen Group (Active Comparator): Patients will be prescribed the current department-wide postoperative pain protocol as described in the Intervention Description.
  Interventions: Drug: Standard of Care Pain Regimen
- Multimodal Pain Regimen Group (Experimental): Multimodal pain regimen medications will be prescribed and administered preoperatively in preoperative holding area, intraoperatively during the procedure, and postoperatively as described in the Intervention Description.
  Interventions: Drug: Multimodal Pain Regimen

INTERVENTIONS:
Drug: Multimodal Pain Regimen — Preoperatively: One dose of Pregabalin 100mg and Celecoxib 400mg along with interscalene block
  Intraoperatively: Intravenous Dexamethasone 0.1mg/kg (maximum dose of 8mg), Magnesium 2g, Acetaminophen 1000mg, and local infiltration of 0.5% Ropivacaine 20ml
  Postoperatively (Discharge): Acetaminophen 975mg every 4 hours, Meloxicam 7.5mg once per day, Pregabalin 50mg twice per day, Magnesium 400mg once per day, along with rescue Oxycodone 5mg every 4 hours, as needed
  Arms: Multimodal Pain Regimen Group
Drug: Standard of Care Pain Regimen — No preoperative medications. Interscalene block in the preoperative holding area. Alternating Acetaminophen 975mg and Ibuprofen 600mg every 4 hours, with rescue Oxycodone 5mg every 4 hours, as needed
  Arms: Standard Pain Regimen Group

SUMMARY:
The goal of this clinical trial is to understand which group of pain control medications work best in adults after rotator cuff surgery.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether a previously described multimodal pain protocol involving non-narcotic medications compared to the medical center's current postoperative pain regimen mainly involving narcotics will decrease total rescue narcotics used for patients who undergo arthroscopic rotator cuff tear repair at Montefiore. The implications of the study would be reduced narcotics consumptions in postoperative patients and improved self-reported patient outcomes. Through this study, the investigator team hopes to develop a pain regimen that alleviates dependence on opioids in postoperative patients without sacrificing patient satisfaction and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Adults with rotator cuff tears who have failed conservative therapy and are now undergoing arthroscopic rotator cuff repair.

Exclusion Criteria:

* Patients without capacity to consent for the study
* Patients not able to have local nerve block
* Patients who underwent previous shoulder surgery on the same side, kindling revision rotator cuff repair
* Patients who are unable to record and verbalize their pain level due to altered mental status
* Patients who are unable to tolerate any of the medications included in the multimodal pain regimen or standard pain regimen due to severe allergies or inability to consume medication
* Patients with history of previously diagnosed alcohol or drug abuse, renal impairment, peptic ulcer disease, and gastrointestinal bleeding
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative narcotics usage | Post-operative day 7
  Post-operative narcotics usage will be assessed by the number of oxycodone tablets used in the first week (7 days) after surgery. The week's use will be accounted by counting the left-over oxycodone tablets brought in by the patients. In addition, the electronic medical record will be checked to ensure that no extra narcotics were called in. Results will be summarized by study arm using means and standard deviations.
Pain Score using the Visual Analogue Scale (VAS) | Post-operative day 7
  A pain score will be determined using the VAS, a unidimensional measure of pain intensity. Patients will be asked to rate and record pain intensity daily during the study. The VAS score at post-operative day 7 will be reported. The VAS score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100, such that higher scores are indicative of greater pain intensity. Results will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Chan, M.D., Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Hutchinson Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones MR, Viswanath O, Peck J, Kaye AD, Gill JS, Simopoulos TT. A Brief History of the Opioid Epidemic and Strategies for Pain Medicine. Pain Ther. 2018 Jun;7(1):13-21. doi: 10.1007/s40122-018-0097-6. Epub 2018 Apr 24. PMID 29691801
- [Background] Storesund A, Krukhaug Y, Olsen MV, Rygh LJ, Nilsen RM, Norekval TM. Females report higher postoperative pain scores than males after ankle surgery. Scand J Pain. 2016 Jul;12:85-93. doi: 10.1016/j.sjpain.2016.05.001. Epub 2016 May 27. PMID 28850501
- [Background] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Background] Moutzouros V, Jildeh TR, Khalil LS, Schwartz K, Hasan L, Matar RN, Okoroha KR. A Multimodal Protocol to Diminish Pain Following Common Orthopedic Sports Procedures: Can We Eliminate Postoperative Opioids? Arthroscopy. 2020 Aug;36(8):2249-2257. doi: 10.1016/j.arthro.2020.04.018. Epub 2020 Apr 28. PMID 32353620